CLINICAL TRIAL: NCT04600947
Title: A Multicenter, Open-Label, Single-arm Phase II Study of LP002 in Subjects With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma
Brief Title: Study of LP002 for the Treatment of Patients With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taizhou HoudeAoke Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP002-II-PMBL-01
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Primary Mediastinal Large B-Cell Lymphoma (PMBCL)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LP002 (Experimental): Participants will receive LP002 10 mg/kg by intravenous (IV) infusion every 2 weeks (Q2W) for up to 24 months.
  Interventions: Drug: LP002

INTERVENTIONS:
Drug: LP002 — 10 mg/kg administered as IV infusion on Day 1 of each 14-day cycle.

SUMMARY:
LP002 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors. In this study, the efficacy and safety of LP002 for the treatment of relapsed or refractory primary mediastinal large B-cell lymphoma will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial;
2. Age ≥ 18 years old, male or female;
3. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score;
4. Life expectancy ≥ 3 months;
5. Subjects must have histopathological diagnosis of primary mediastinal large B-cell lymphoma (PMBCL), according to the WHO classification of lymphoma (revised in 2017) (diagnosis is confirmed by the central pathological review), and meet the following criteria:

   1. Recurrence after autologous hematopoietic stem cell transplantation (ASCT), or complete remission (CR) or partial remission (PR) is not achieved within 60 days after ASCT. If patients with relapse or refractory ASCT receive other interventions, they must be relapsed or refractory after the last systemic treatment;
   2. Patients who are not suitable for ASCT must be second-line or above chemotherapy invalid or recurring; local radiotherapy alone is not considered as first-line treatment;
   3. Need to be treated with rituximab, or cannot be treated with rituximab for any reason;
6. According to the Lugano standard in 2014, CT/MRI should show that there is at least one measurable tumor lesion in two vertical directions, with the length of the intranodal lesion ≥1.5cm and the length of the extranodal lesion ≥1.0cm;
7. The subject has sufficient organ and bone marrow function to meet the following laboratory examination standards:

   1. Blood routine: absolute neutrophil count (ANC)≥1.0×10^9/L; platelet count (PLT)≥80×10^9/L; hemoglobin (HGB)≥8.0 g/dL; Note: It is not allowed to use any blood components, cell growth factors and other interventions within 14 days before the examination.
   2. Liver function: Patients without liver metastases require serum total bilirubin (TBIL) ≤1.5×upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN. Patients with liver metastases require: TBIL≤1.5×ULN; ALT and AST≤5×ULN;
   3. Renal function: Serum creatinine (Scr) ≤1.5×ULN, or endogenous creatinine clearance ≥50 mL/min (Cockcroft-Gault formula);
   4. The coagulation function is adequate, which is defined as the international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 times ULN;
8. Reproductive men and women of childbearing age are willing to take effective contraceptive measures from signing the informed consent form to 6 months after the last administration of the trial drug. Women of childbearing age must have a negative blood pregnancy test within 7 days before the first trial drug administration.

Exclusion Criteria:

1. Suffered from other malignant tumors in the past 3 years (except skin basal cell carcinoma, squamous cell carcinoma, and cervical carcinoma in situ that have been effectively controlled);
2. Currently participating in interventional clinical research treatment, or receiving other experimental drugs or using experimental device treatment within 4 weeks before the first administration;
3. Received systemic systemic chemotherapy or targeted drug therapy within 4 weeks or 5 half-lives before the first administration;
4. The study drug has received anti-tumor indications Chinese herbal medicine, or immunomodulatory drugs (including thymosin, interferon, interleukin, etc., except for local use to control pleural effusion or pericardial effusion) within 2 weeks before the first administration Systemic systemic therapy;
5. Received monoclonal antibody drug treatment within 4 weeks before the first administration;
6. Received radical or palliative radiotherapy within 4 weeks before the first administration;
7. Received autologous stem cell transplantation within 8 weeks before the first administration;
8. Prior to the first administration of the study drug, there was a grade > 1 toxicity (excluding hair loss, non-clinical) caused by previous anti-tumor treatments;
9. Previously used anti-PD-1, anti-PD-L1, anti-programmed cell death protein ligand 2 (PD-L2) or anti-cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) drugs or acted on T cell co-stimulation Or any other drugs in the checkpoint pathway;
10. Have received systemic corticosteroids or other immunosuppressive drugs within 2 weeks before the first administration of the study drug, excluding:

    1. Nasal spray, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (ie ≤10mg/day prednisone or its equivalent dose of other glucocorticoids);
    2. Short-term use of glucocorticoids as a preventive medication for allergic reactions (such as prevention of contrast agent allergy);
    3. Short-term use of glucocorticoids to treat non-autoimmune diseases (such as delayed type hypersensitivity caused by contact allergens);
11. Has central nervous system (CNS) invasion, including brain parenchyma, meningeal invasion, or spinal cord compression;
12. A history of active and known autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel disease, Hashimoto's thyroiditis, etc., except: Type I Diabetes, hypothyroidism that can be controlled only by hormone replacement therapy, skin diseases that do not require systemic treatment (such as vitiligo, psoriasis), controlled celiac disease, or diseases that are not expected to recur without external stimuli;
13. Has a history of or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severely impaired lung function and other lung diseases;
14. Severe chronic or active infections that require systemic antibacterial, antifungal or antiviral therapy, including tuberculosis, syphilis (TP-Ab positive), AIDS (HIV antibody positive), etc.;
15. Known history of human immunodeficiency virus (HIV) infection; acute or chronic active hepatitis B (HBsAg positive and HBV DNA viral load ≥200 IU/mL or ≥10^3 copies/mL); acute or chronic active Hepatitis C (HCV antibody positive and HCV RNA positive);
16. Within 4 weeks before the first administration of the study drug or plan to receive live vaccines or live attenuated vaccines during the study period;
17. Has received a major surgical operation within 4 weeks before the first treatment with the study drug or is expected to undergo major surgery during the study treatment;
18. Known to be allergic to recombinant humanized PD-L1 monoclonal antibody or any of its excipients; Known to have a history of allergic diseases or have severe allergies;
19. Cardiovascular diseases meet any of the following: congestive heart failure with heart function ≥ NYHA II; severe arrhythmia requiring medical treatment; acute myocardial infarction, severe or unstable angina pectoris occurred within 6 months before the first administration, coronary or peripheral artery bypass, stenting; left ventricular ejection fraction (LVEF) <50%; corrected QTcF interval> 450 milliseconds for men and> 470 milliseconds for women, or there is a risk of torsade de pointes ventricular tachycardia factors such as clinically significant hypokalemia, family history of long QT syndrome, or family history of arrhythmia (such as pre-excitation syndrome) as judged by the investigator; hypertension that cannot be effectively controlled (defined as standardized antihypertensive drugs after treatment, systolic blood pressure ≥140 mmHg and/or diastolic blood pressure >90 mmHg);
20. Pleural fluid, ascites, and pericardial effusion with clinical symptoms requiring drainage;
21. Combined with other serious medical diseases, including but not limited to: uncontrolled diabetes, active peptic ulcer, active bleeding, etc.;
22. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.
23. According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 24 months
  Percentage of subjects achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | up to approximately 24 months
  Progression-free survival (PFS) is defined as the time from the first study drug treatment to disease progression (PD) or to death of the subject due to any reason. For subjects whose progression or death is unknown, PFS will be censored at the time of the last valid evaluation.
Duration of Response (DOR) | up to approximately 24 months
  Duration of Response (DOR) is defined as the time from the first evidence of repsonse (PR or CR) to the first evidence of PD or the date of death for any reason in patients who have been confirmed to have response (2014 Lugano criteria, PR or CR).
Time to Response (TTR) | up to approximately 24 months
  Time to Response (TTR) refers to the time from the first treatment with the study drug to the first CR or PR on tumor evaluation.
Disease Control Rate (DCR) | up to approximately 24 months
  Disease Control Rate (DCR) refers to the proportion of subjects who achieve CR, PR and SD through imaging evaluation.
Overall survival (OS) | up to approximately 24 months
  Overall survival (OS) refers to the time from the first study drug treatment to death due to any cause. For subjects who have not been followed up to death, OS will be censored at the last effective survival follow-up time.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (7):
- China (7):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan